CLINICAL TRIAL: NCT01021319
Title: PREdictive Value of FLAIR and DWI for the Identification of Acute Ischemic Stroke Patients ≤ 3 and ≤ 4.5 h of Symptom Onset - a Multicenter Observational Study
Brief Title: Identification of Stroke Patients ≤ 3 and ≤ 4.5 Hours of Symptom Onset by Fluid Attenuated Inversion Recovery (FLAIR) Imaging and Diffusion Weighted Imaging (DWI)
Acronym: PRE-FLAIR
Status: Completed | Type: Observational
Sponsor: Götz Thomalla, MD (Other)
Collaborators: Else Kröner-Fresenius-Stiftung (Foundation) (Unknown); Stroke Imaging Repositoy (STIR) (Unknown); MR Stroke Group (Unknown)
Responsible Party: Sponsor-Investigator, Götz Thomalla, MD, PD Dr. med. Götz Thomalla, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: PRE-FLAIR
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Ischemic Stroke
Keywords: ischemic stroke; thrombolysis; magnetic resonance imaging; diffusion weighted imaging; fluid attenuated inversion recovery; time window
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute ischemic stroke: Patients with acute ischemic stroke confirmed by acute or follow-up MRI with defined andwell-known symptom onset.

SUMMARY:
The aim of the study is to evaluate the use of combined fluid attenuated inversion recovery (FLAIR) imaging and diffusion weighted imaging (DWI) as surrogate marker of lesion age within the first 6 hours of ischemic stroke in order to identify patients ≤ 3 or ≤ 4.5 hours of symptom onset in a large multicenter study hours of ischemic stroke. The investigators hypothesize that the pattern of a visible lesion on DWI together with a negative FLAIR ("DWI-FLAIR mismatch") will identify patients ≤ 3 hours of symptom onset with >80% specificity and positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke (proven by initial or follow-up MRI)
* Well defined and known symptom onset
* Stroke MRI including diffusion weighted imaging (DWI) and fluid attenuated inversion recovery (FLAIR) sequences performed within 12 hours of symptom onset
* Informed consent

Exclusion Criteria:

* Contraindications against MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke confirmed by acute or follow-up MRI with defined and well known symptom onset
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Specificity (and 95% CI) of "DWI-FLAIR-mismatch" for the identification of patients ≤3 and ≤4.5 hours | on admission

SECONDARY OUTCOMES:
Predictors of a "negative FLAIR" in acute ischemic stroke | on admission

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, MD, Principal Investigator — Uinversity Medical Center Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Charite Clinical Center, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Result] Thomalla G, Cheng B, Ebinger M, Hao Q, Tourdias T, Wu O, Kim JS, Breuer L, Singer OC, Warach S, Christensen S, Treszl A, Forkert ND, Galinovic I, Rosenkranz M, Engelhorn T, Kohrmann M, Endres M, Kang DW, Dousset V, Sorensen AG, Liebeskind DS, Fiebach JB, Fiehler J, Gerloff C; STIR and VISTA Imaging Investigators. DWI-FLAIR mismatch for the identification of patients with acute ischaemic stroke within 4.5 h of symptom onset (PRE-FLAIR): a multicentre observational study. Lancet Neurol. 2011 Nov;10(11):978-86. doi: 10.1016/S1474-4422(11)70192-2. Epub 2011 Oct 4. PMID 21978972